CLINICAL TRIAL: NCT02358928
Title: Low Carbohydrate Diet: The Effects on Non Alcoholic Fatty Liver Disease in Obese Teens With Metabolic Syndrome
Acronym: NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Charina Ramirez, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 082013 020
Record Dates: First submitted 2015-01-29; First posted 2015-02-09 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: NAFLD; Fatty Liver; Obesity; Metabolic Syndrome
Keywords: NAFLD; Metabolic syndrome; Hepatic Magnetic Resonance Spectroscopy; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low calorie diet (Other): Calorie-restricted diet is composed of 50% carbohydrate, 15-20% protein and 30-35% fat.
  Interventions: Other: Diet Intervention
- Low carbohydrate diet (Other): Carbohydrate-restricted diet is composed of 20% carbohydrates, 35% protein and 45% fat.
  Interventions: Other: Diet Intervention

INTERVENTIONS:
Other: Diet Intervention

SUMMARY:
Concurrent with the rising prevalence of childhood obesity, the co-morbid condition of non-alcoholic fatty liver disease (NAFLD) has become the leading cause of chronic liver disease among children. NAFLD is characterized by accrual of excess triglycerides (TG) in the liver that leads to inflammation, fibrosis, and cirrhosis. One-third of the pediatric population has NAFLD, a disease strongly associated with insulin-resistance and metabolic-syndrome (Met-S). NAFLD is predicted to become the leading cause of liver transplantation in adults by 2030.

Current understanding of NAFLD indicates that presence of excess TG in liver is an absolute requirement for disease progression. First-line therapy for NAFLD is focused on decreasing adiposity and improving insulin sensitivity through diet and exercise. Recent adult data indicate that dietary carbohydrate-restriction is more effective at reducing hepatic TG-content than traditional calorie-restriction. Few studies have been conducted to establish resolution of hepatic steatosis by any intervention. Such studies in pediatrics are primarily limited by a need for liver biopsy. However, hepatic proton magnetic resonance spectroscopy (H-MRS) is a new innovative tool used to quantitatively measure hepatic TG content in a non-invasive manner.

The primary aim is to compare the impact of dietary weight loss via carbohydrate-restriction and calorie-restriction on hepatic TG-content quantified by H-MRS in obese children with biopsy-proven NAFLD and Met-S.

This IRB approved protocol is a randomized control study. The investigators will recruit subjects from the Center for Obesity and its Consequences in Health and the pediatric gastroenterology clinics between the ages of 11-17 years who meet criteria for NAFLD and Met-S. A H-MRS will be obtained in each subject prior to the start of dietary intervention. Fifty-four subjects will be randomized to either a carbohydrate-restricted or calorie-restricted diet for 6 months with no change in baseline activity. A repeat H-MRS will be compared to baseline to determine the whether dietary carbohydrate-restriction is superior to calorie-restriction for reducing hepatic TG content. The investigators believe that subjects on the carbohydrate-restricted diet will have marked decrease in hepatic TG content compared to those in the calorie-restricted diet given the same degree of reduction in body mass index.

DETAILED DESCRIPTION:
Specific Aims and Hypothesis:

The Primary aim is:

To compare the impact of dietary weight loss via carbohydrate-restriction and calorie-restriction on hepatic TG content quantified by H-MRS in obese children with biopsy-proven NAFLD and Met-S.

Our Secondary aims are:

To compare BMI z-score, ALT (analine transaminase) and cytokeratin 18 in obese patients with NAFLD and Met-S after a 6 month dietary weight loss via either carbohydrate or calorie restriction.

Hypothesis: Obese children with biopsy-proven NAFLD and Met-S will experience a reduction in liver TG content, assessed by H-MRS, concurrent with 6 months of dietary weight loss; however, we anticipate that subjects undergoing carbohydrate restriction will experience a greater reduction in hepatic fat than those undergoing calorie restriction due to the limiting of precursors for lipid synthesis inherent to the diet (CHO) and the expected increase in hepatic oxidative metabolism (TG accrual is attenuated while disposal is enhanced).

Methodology:

Design:

Our study is a 6 month prospective randomized controlled trial with outcomes assessment monthly for the first 6 months and a follow up visit at 10- 12 months after randomization.

Setting:

Recruitment and data collection will be completed at University of Texas Southwestern Medical Center and Children's Health, Dallas TX by study personnel. All patients who agree to participate will give informed written consent and assent. A study staff member will explain the study and review the consent and HIPAA forms with each patient. A copy of each signed form will be kept in the patient's study file. Each patient will also receive signed copies.

Subjects:

All patients referred (male and female) within the age range of 11 - 17 years who are obese (BMI >= 95th percentile) and meet criteria for metabolic syndrome (MetS) and non-alcoholic fatty liver disease (NAFLD) will be offered to participate in study.

Inclusion Criteria:

1. Age 11 - 17 years
2. Male and Female subjects
3. BMI >= 95th percentile according to CDC body mass index chart for age and gender
4. Must be willing to participate and undergo "willingness to change" evaluation
5. Metabolic Syndrome(MetS) which is defined when 3 of the following are met:

   1. Central adiposity (waist circumference ≥90th% for age and sex)
   2. Hypertriglyceridemia (triglycerides ≥ 110mg/dl)
   3. Low HDL cholesterol ≤40mg/dl
   4. Elevated blood pressure systolic or diastolic blood pressure > 90th % adjusted for age, sex and height or ≥ 130/85
   5. IFG (Impaired fasting glucose ≥ 100mg/dl or elevated HOMA- IR ≥3.16)
6. ALT greater than 60 U/L and Non Alcoholic Fatty Liver Disease based on histologic confirmation on liver biopsy (minimum of 5% of hepatocytes with macrovesicular fat) obtained within 6 months before randomization

Exclusion Criteria:

1. Those patients with a history of poor compliance or adherence to energy restriction diets
2. Patients on medications that could alter appetite including glucocorticoids, psychostimulants (Vyvanse, Adderall), psychotropic medications (Zoloft, Risperdal), and antihyperglycemic medications (metformin, sulfonylurea)
3. Patients with the following illnesses:

   1. Type 2 diabetes
   2. Renal disease
   3. Mental diseases (mood, psychotic and anxiety disorders)
   4. Developmental delay
   5. Autism and autism spectrum disorders
   6. Any liver disease except for non alcoholic fatty liver (NAFLD)
   7. Metabolic disorders (tyrosinemia, glycogen storage disease, lysosomal disorders)
   8. Congenital heart disease
   9. Myopathies or muscular disorders/disability
4. Patients who follow a (cultural or religious) vegetarian lifestyle as this would not be compatible with Carbohydrate Restriction (need for high quality protein)
5. Prepubertal patients defined by a tanner stage of 1
6. Current or history of significant alcohol consumption

Concise Summary of Project:

This is a 6-month prospective, randomized control trial enrolling patients referred to the Children's Medical Center COACH Program. The COACH Program is a medical weight management clinic, which serves obese children in order to diagnose and treat associated co-morbid conditions.

Subjects meeting all enrollment criteria will be randomized to either a carbohydrate- or calorie-restricted diet. They will be committed to this fixed meal plan for 6 months and dietary education by a certified dietician will be provided. This will include the allowed caloric intake and content, which is calculated by a bioelectric impedance meter (GE In Body 520) specific to patient's age, gender, and weight.

The carbohydrate-restricted diet is composed of 20% carbohydrates, 35% protein and 45% fat. The calorie-restricted diet is composed of 50%carbohydrate, 15-20% protein and 30-35% fat. Patients will be seen by a psychologist to help with goal setting, self-monitoring and problem solving. Dietary compliance will be followed regularly by weekly phone calls for the first 3 months and then monthly afterwards by the research personnel. A 72-hour dietary recall will be conducted by our dietician every other month. Subjects will be followed in the COACH clinic monthly. A detailed schedule will be outlined and provided to the families at each visit. Any missed appointments will be rescheduled within 3 to 7 days, and the families will be contacted immediately to offer assistance for the next visit. During this study, subjects will be monitored with urine tests and blood tests to ensure safety while undergoing the prescribed diet.

The first proton hepatic magnetic spectroscopy (H-MRS) will be done prior to initiating the dietary intervention. A second H-MRS will be obtained after 2 months (at visit 3) on the assigned dietary therapy. The final H-MRS will be performed after completion of the 6 month dietary intervention. At the 6 month completion, the subjects will be seen in clinic and blood work with urine testing will be done. Their final visit will be 4 to 6 months post dietary intervention to assess weight maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 11 - 17 years
2. Male and Female subjects
3. BMI >= 95th percentile according to CDC body mass index chart for age and gender
4. Must be willing to participate and undergo "willingness to change" evaluation
5. Metabolic Syndrome(MetS) which is defined when 3 of the following are met:

   * Central adiposity (waist circumference ≥90th% for age and sex)
   * Hypertriglyceridemia (triglycerides ≥ 110mg/dl)
   * Low HDL cholesterol ≤40mg/dl
   * Elevated blood pressure systolic or diastolic blood pressure > 90th % adjusted for age, sex and height or ≥ 130/85
   * IFG (Impaired fasting glucose ≥ 100mg/dl or elevated HOMA- IR ≥3.16)
6. ALT greater than 60 U/L and Non Alcoholic Fatty Liver Disease based on histologic confirmation on liver biopsy (minimum of 5% of hepatocytes with macrovesicular fat) obtained within 6 months before randomization

Exclusion Criteria:

1. Those patients with a history of poor compliance or adherence to energy restriction diets
2. Patients on medications that could alter appetite including glucocorticoids, psychostimulants (Vyvanse, Adderall), psychotropic medications (Zoloft, Risperdal), and antihyperglycemic medications (metformin, sulfonylurea)
3. Patients with the following illnesses:

   * Type 2 diabetes
   * Renal disease
   * Mental diseases (mood, psychotic and anxiety disorders)
   * Developmental delay
   * Autism and autism spectrum disorders
   * Any liver disease except for non alcoholic fatty liver (NAFLD)
   * Metabolic disorders (tyrosinemia, glycogen storage disease, lysosomal disorders)
   * Congenital heart disease
   * Myopathies or muscular disorders/disability
4. Patients who follow a (cultural or religious) vegetarian lifestyle as this would not be compatible with Carbohydrate Restriction (need for high quality protein)
5. Prepubertal patients defined by a tanner stage of 1
6. Current or history of significant alcohol consumption

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

PRIMARY OUTCOMES:
HepaticTrigylceride Content quantified on proton magnetic spectroscopy (H-MRS) | 1 year
  To compare the impact of dietary weight loss via carbohydrate-restriction and calorie-restriction on hepatic TG content quantified by H-MRS in obese children with biopsy-proven NAFLD and Met-S.

SECONDARY OUTCOMES:
BMI Z-score | 1 year
  To compare BMI z-score in obese patients with NAFLD and Met-S after a 6 month dietary weight loss via either carbohydrate or calorie restriction.
Cytokeratin-18 | 1 year
  Quantify the effect of dietary weight loss via carbohydrate- and calorie-restriction on serum markers of hepatic fibrosis.
ALT (alanine transaminase) | 1 year
  To compare ALT in obese patients with NAFLD and Met-S after a 6 month dietary weight loss via either carbohydrate or calorie restriction.

CONTACTS AND LOCATIONS:
Overall Officials: Charina Ramirez, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UTexasSouthwestern/Childrens Medical Center, Dallas, Texas, United States